CLINICAL TRIAL: NCT03657797
Title: A Phase 2, Randomized, Multicenter, Masked, Parrallel-Group, Dose-Response Study Evaluating the Safety and Efficacy of NCX 470 (3 Doses: 0.021%, 0.042%, and 0.065%) vs. Latanoprost 0.005% in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Phase 2 Dose-Response Study Evaluating the Safety and Efficacy of NCX 470 vs Latanoprost in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nicox Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCX-470-17001
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Results first posted 2022-12-08 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Glaucoma, Open-Angle; Hypertension, Ocular
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NCX 470 0.021% (Experimental): NCX 470 Ophthalmic Solution, 0.021% dosed once daily for 4 weeks
  Interventions: Drug: NCX 470
- NCX 470 0.042% (Experimental): NCX 470 Ophthalmic Solution, 0.042% dosed once daily for 4 weeks
  Interventions: Drug: NCX 470
- NCX 470 0.065% (Experimental): NCX 470 Ophthalmic Solution, 0.065% dosed once daily for 4 weeks
  Interventions: Drug: NCX 470
- Latanoprost 0.005% (Active Comparator): Latanoprost Ophthalmic Solution, 0.005% dosed once daily for 4 weeks
  Interventions: Drug: Latanoprost 0.005%

INTERVENTIONS:
Drug: NCX 470 — NCX 470 Ophthalmic Solution
  Arms: NCX 470 0.021%; NCX 470 0.042%; NCX 470 0.065%
Drug: Latanoprost 0.005% — Latanoprost 0.005% Ophthalmic Solution
  Other Names: Latanoprost
  Arms: Latanoprost 0.005%

SUMMARY:
The objective of this clinical study is to evaluate the safety and efficacy of NCX 470 ophthalmic solution in lowering intraocular pressure (IOP) in patients with ocular hypertension or open-angle glaucoma. Three different concentrations of NCX 470 ophthalmic solution (0.021%, 0.042%, and 0.065%) will be compared to latanoprost 0.005% ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension in both eyes
* Qualifying IOP at 3 time points throughout the day at 2 visits following washout of IOP-lowering medication, if applicable
* Qualifying best-corrected visual acuity (BCVA) using the Early Treatment of Diabetic Retinopathy Study (ETDRS) protocol in each eye
* Ability to provide informed consent and follow study instructions

Exclusion Criteria:

* Pigmentary or pseudoexfoliative glaucoma
* Narrow anterior chamber angles or disqualifying corneal thickness in either eye
* Clinically significant ocular disease in either eye
* Previous complicated surgery or certain types of glaucoma surgery in either eye
* Incisional ocular surgery or severe trauma in either eye within the past 6 months
* Uncontrolled systemic disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicox Ophthalmics, Inc., Study Director — Nicox Ophthalmics, Inc.
Locations (1):
- Texan Eye, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ophthalmologists' clinics in the US. The first participant for the study was screened in August 2018 and the last participant exited the trial in August 2019.
Pre-assignment Details: Potential participants were screened for eligibility and those on intraocular pressure (IOP) lowering medication were required to undergo a wash out of 5 to 42 days (dependent on the class of medication). After the appropriate washout period, or after a minimum of 5 days for participants who were not on IOP lowering medication at screening, participants underwent 2 eligibility visits held 3 to 7 days apart. Those who qualified were randomized to one of the 4 treatment groups.
Units Other Than Participants: study eyes
Period: Overall Study
Arm/Group | NCX 470 0.021% | NCX 470 0.042% | NCX 470 0.065% | Latanoprost 0.005%
Started | 111; 111 study eyes (Met inclusion/exclusion criteria, including IOP entry criteria at 2 eligibility visits) | 108; 108 study eyes (Met inclusion/exclusion criteria, including IOP entry criteria at 2 eligibility visits) | 107; 107 study eyes (Met inclusion/exclusion criteria, including IOP entry criteria at 2 eligibility visits) | 107; 107 study eyes (Met inclusion/exclusion criteria, including IOP entry criteria at 2 eligibility visits)
Completed | 111; 111 study eyes | 105; 105 study eyes | 102; 102 study eyes | 107; 107 study eyes
Not Completed | 0; 0 study eyes | 3; 3 study eyes | 5; 5 study eyes | 0; 0 study eyes
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants contribute a study eye (fellow eye also treated)
Groups:
- Total: Total of all reporting groups
Arm/Group | NCX 470 0.021% | NCX 470 0.042% | NCX 470 0.065% | Latanoprost 0.005% | Total
Number analyzed (Participants) | 111 | 108 | 107 | 107 | 433
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 46 | 53 | 55 | 202
  >=65 years | 63 | 62 | 54 | 52 | 231
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 71 | 58 | 57 | 240
  Male | 57 | 37 | 49 | 50 | 193
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 20 | 16 | 18 | 77
  Not Hispanic or Latino | 88 | 88 | 91 | 89 | 356
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 2 | 1 | 3 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 35 | 32 | 32 | 35 | 134
  White | 72 | 74 | 71 | 70 | 287
  More than one race | 2 | 1 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 111 | 108 | 107 | 107 | 433
Study Eye Baseline Mean Diurnal IOP (mmHg) [Mean (Standard Deviation); unit: mmHg] — Average of study eye IOP measured at 8AM,10AM and 4PM at 2 eligibility visits
  mmHg | 26.62 (1.663) | 26.89 (1.987) | 26.80 (2.069) | 26.68 (1.745) | 26.75 (1.866)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Study Eye Mean Diurnal IOP at the Week 4
Description: Participants used medication in both eyes for 4 weeks with one eye was designated the study eye at baseline. The study eye was defined as the eye with the highest mean diurnal intraocular pressure (IOP) value at baseline (or the right eye if both eyes had the same IOP value at baseline). Mean diurnal IOP at week 4 is the average of the 8AM, 10AM and 4PM IOPs at week 4.
Time Frame: Baseline, Week 4
Population: All participants who were randomized and who had diurnal IOP values at week 4
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: study eyes
Groups:
- NCX 470 0.021%: Participants received NCX 470 0.021% once daily in both eyes
- NCX 470 0.042%: Participants received NCX 470 0.042% once daily in both eyes
- NCX 470 0.065%: Participants received NCX 470 0.065% once daily in both eyes
- Latanoprost 0.005%: Participants received latanoprost 0.005% once daily in both eyes
Arm/Group | NCX 470 0.021% | NCX 470 0.042% | NCX 470 0.065% | Latanoprost 0.005%
Number analyzed (Participants) | 110 | 105 | 102 | 107
Number analyzed (study eyes) | 110 | 105 | 102 | 107
mmHg | -7.79 (2.606) | -8.28 (2.511) | -8.70 (3.150) | -7.41 (2.666)
Statistical Analysis 1: Comparison: NCX 470 0.021% vs Latanoprost 0.005%; NCX 470 0.21% was compared to latanoprost; Test type: Non-Inferiority — LS mean, the difference in LS mean (NCX 470 minus latanoprost), and the 2-sided 95% CI for the difference was obtained. Non-inferiority could be claimed if the upper limit of the 2-sided 95% CI around the difference between the LS mean for NCX 470 and the LS mean for latanoprost was < 1.5 mmHg. If non-inferiority was met, superiority was tested which could be claimed if the p-value for treatment difference was <= 0.05 and the LS mean difference in change from baseline was < 0; p = 0.2666, ANCOVA — p-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-1.11 to 0.31]
Statistical Analysis 2: Comparison: NCX 470 0.042% vs Latanoprost 0.005%; NCX 0.042% was compared to latanoprost; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0281, ANCOVA — p-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.52 to -0.09]
Statistical Analysis 3: Comparison: NCX 470 0.065% vs Latanoprost 0.005%; NCX 0.065% was compared to latanoprost; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0009, ANCOVA — p-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-1.96 to -0.51]

2. Secondary Outcome: Change From Baseline in Study Eye Mean Diurnal IOP at Week 1, Week 2, and Exit Visit
Description: Participants used medication in both eyes from baseline to the evening prior to the week 4 visit. One eye was designated the study eye at baseline. The study eye was defined as the eye with the highest mean diurnal intraocular pressure (IOP) value at baseline (or the right eye if both eyes had the same IOP value at baseline). Mean diurnal IOP is the average of the 8AM, 10AM and 4PM values. Visits were conducted at week 1, week 2, week 4, and an exit visit (1 to 2 days following the week 4 visit)
Time Frame: Baseline, week 1, week 2, exit visit
Population: All participants who were randomized and who had diurnal IOP values at the week 1, week 2, exit visits
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: study eyes
Arm/Group | NCX 470 0.021% | NCX 470 0.042% | NCX 470 0.065% | Latanoprost 0.005%
Number analyzed (Participants) | 111 | 108 | 107 | 107
Number analyzed (study eyes) | 111 | 108 | 107 | 107
mmHg
  Week 1: number analyzed (Participants) | 110 | 108 | 104 | 107
  Week 1: number analyzed (study eyes) | 110 | 108 | 104 | 107
  Week 1 | -7.73 (2.783) | -8.15 (2.577) | -8.66 (3.098) | -7.54 (2.735)
  Week 2: number analyzed (Participants) | 111 | 106 | 104 | 107
  Week 2: number analyzed (study eyes) | 111 | 106 | 104 | 107
  Week 2 | -7.96 (2.774) | -8.38 (2.439) | -8.87 (2.797) | -7.99 (2.504)
  Exit Visit: number analyzed (Participants) | 110 | 105 | 102 | 106
  Exit Visit: number analyzed (study eyes) | 110 | 105 | 102 | 106
  Exit Visit | -4.95 (3.237) | -5.59 (2.827) | -5.98 (3.019) | -4.89 (3.009)
Statistical Analysis 1: Comparison: NCX 470 0.021% vs Latanoprost 0.005%; NCX 470 0.021% was compared to latanoprost; Test type: Non-Inferiority — NCX 470 0.021% was compared to latanoprost 0.005% at each visit. The LS mean, LS mean difference and the 95% CIs for the difference was calculated. Non-inferiority at each visit could be claimed if the upper limit of the 95% CI was <1.5 mmHg. If non-inferiority was established, superiority could be claimed if the upper limit of the 95% CI was <0 and p<0.05; p < 0.9788, ANCOVA — p-value was not adjusted for multiple comparisons; Upper 95% CIs were 0.51 (week 1), 0.68 (week 2), 0.75 (exit visit); p-values were 0.5560 (week 1), 0.9788 (week 2), 0.8796 (exit visit)
Statistical Analysis 2: Comparison: NCX 470 0.042% vs Latanoprost 0.005%; NCX 470 0.042% was compared to latanoprost; Test type: Non-Inferiority — NCX 470 0.042% was compared to latanoprost 0.005% at each visit. The LS mean, LS mean difference and the 95% CIs for the difference was calculated. Non-inferiority at each visit could be claimed if the upper limit of the 95% CI was <1.5 mmHg. If non-inferiority was established, superiority could be claimed if the upper limit of the 95% CI was <0 and p<0.05; p < 0.3863, ANCOVA — p-value was not adjusted for multiple comparisons; Upper 95% CIs were 0.20 (week 1), 0.38 (week 2), 0.11 (exit visit); p-values were 0.1556 (week 1), 0.3863 (week 2), 0.0912 (exit visit)
Statistical Analysis 3: Comparison: NCX 470 0.065% vs Latanoprost 0.005%; NCX 470 0.065% was compared to latanoprost; Test type: Non-Inferiority — NCX 470 0.065% was compared to latanoprost 0.005% at each visit. The LS mean, LS mean difference and the 95% CIs for the difference was calculated. Non-inferiority at each visit could be claimed if the upper limit of the 95% CI was <1.5 mmHg. If non-inferiority was established, superiority could be claimed if the upper limit of the 95% CI was <0 and p<0.05; p < 0.0174, ANCOVA — p-value was not adjusted for multiple comparisons; Upper 95% CIs were -0.35 (week 1), -0.15 (week 2), -0.27 (exit visit); p-values were 0.0040 (week 1), 0.0174 (week 2), 0.0093 (exit visit)

3. Secondary Outcome: Percentage of Subjects With Treatment-emergent Ocular Adverse Events
Description: Safety and tolerability based on percentage of subjects with treatment-emergent ocular adverse events
Time Frame: 4 weeks for adverse events and through 30 days post-treatment for serious adverse events
Population: Safety population defined as all participants who received at least one dose of the study medication during the 4-week treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | NCX 470 0.021% | NCX 470 0.042% | NCX 470 0.065% | Latanoprost 0.005%
Number analyzed (Participants) | 111 | 108 | 107 | 107
Participants | 34 | 52 | 50 | 21

ADVERSE EVENTS:
Time Frame: 29 days with collection of serious adverse events for up to 30 days post study exit
Arm/Group | NCX 470 0.021% | NCX 470 0.042% | NCX 470 0.065% | Latanoprost 0.005%
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/108 | 0/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 1/111 | 2/108 | 1/107 | 0/107
Other Adverse Events (participants affected / at risk) | 24/111 | 42/108 | 39/107 | 20/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NCX 470 0.021% (N=111) | NCX 470 0.042% (N=108) | NCX 470 0.065% (N=107) | Latanoprost 0.005% (N=107)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — acute unspecified purulent endophthalmitis following cataract surgery in the 30-day period following completion of study treatment
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Worsening of hypertension
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NCX 470 0.021% (N=111) | NCX 470 0.042% (N=108) | NCX 470 0.065% (N=107) | Latanoprost 0.005% (N=107)
Conjunctival hyperaemia (Eye disorders) | 12 (13) | 24 (25) | 18 (18) | 7 (7)
Ocular hyperaemia (Eye disorders) | 5 (8) | 9 (11) | 10 (12) | 5 (8)
Eye pruritus (Eye disorders) | 2 (2) | 1 (1) | 6 (6) | 0 (0)
Instillation site pain (General disorders) | 8 (8) | 10 (10) | 12 (12) | 6 (6)
Instillation site pruritus (General disorders) | 2 (2) | 5 (5) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT03657797/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT03657797/SAP_001.pdf